CLINICAL TRIAL: NCT00656604
Title: Evaluation of Patients With Breast Cancer Using Dynamic Contrast-Enhanced Magnetic Resonance Imaging, Magnetic Resonance Spectroscopy, and Proteomics
Brief Title: Evaluation of Patients With Breast Cancer Using DCE-MRI, MRS, and Proteomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Associate Professor, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC BRE 0358; P30CA068485 (NIH); VU-VICC-BRE-0358; VU-VICC-IRB-030472
Record Dates: First submitted 2008-04-10; First posted 2008-04-11 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Mastectomy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women with breast cancer (Experimental): Patients undergo DCE-MRI and MRS prior to their breast cancer surgery.
  Interventions: Genetic: proteomic profiling; Procedure: lumpectomy or mastectomy; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: histopathologic examination; Procedure: magnetic resonance spectroscopy
- Healthy volunteers (No Intervention): Women without breast cancer undergo DCE-MRI and MRS.

INTERVENTIONS:
Genetic: proteomic profiling — at the time of each procedure.
  Other Names: proteomic analysis
  Arms: Women with breast cancer
Procedure: lumpectomy or mastectomy — removal of breast tumor or removal of the entire breast in which the tumor is located
  Other Names: None noted
  Arms: Women with breast cancer
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Prior to initiation of treatment
  Other Names: DCE-MRI
  Arms: Women with breast cancer
Procedure: histopathologic examination — After the breast tumor has been removed, examination of the tumor under a microscope to determine the type and grade of breast cancer
  Other Names: Not noted
  Arms: Women with breast cancer
Procedure: magnetic resonance spectroscopy — Prior to initiation of treatment
  Other Names: MRS
  Arms: Women with breast cancer

SUMMARY:
RATIONALE: Diagnostic procedures, such as dynamic contrast-enhanced magnetic resonance imaging(DCE-MRI), magnetic resonance spectroscopy (MRS), and tissue proteomics, may help doctors find and diagnose breast cancer and plan the best treatment.

PURPOSE: This clinical trial is studying MRI and MRS with or without tissue proteomics analysis to see how well they work in evaluating healthy women and women who are undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To correlate data obtained by DCE-MRI and MRS in healthy women and in women who are undergoing surgery for breast cancer with data obtained by conventional X-ray mammography, tissue proteomics, and histopathology.
* To evaluate the impact of MRSI data on treatment planning for radiotherapy and/or surgery.

OUTLINE: Healthy participants undergo dynamic contrast-enhanced (DCE)-MRI and magnetic resonance spectroscopic (MRS) for longitudinal studies of breast imaging and spectroscopy.

Patients with breast cancers undergo DCE-MRI and MRS prior to initiation of treatment (i.e., surgery, chemotherapy, or radiotherapy). After treatment has begun, patients then undergo repeat imaging (not more than 1 per month) for follow-up assessments and longitudinal studies.

Breast tissue samples are collected from patients undergoing surgery. Samples are evaluated by histopathological and proteomic analysis for correlation with DCE-MRI and MRS findings.

The study interventions are discontinued after definitive surgery is performed.

PROJECTED ACCRUAL: A total of 10 healthy participants and 40 patients with breast cancer will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Women with breast tumors planning to undergo surgical resection
  * Healthy volunteers, including any constitutionally healthy female with no history of breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not acutely ill
* No non-magnetic resonance-compatible ferromagnetic materials present in the body

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy and/or radiotherapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Primary Completion 2005-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Correlation of data obtained by DCE-MRI and magnetic resonance spectroscopy (MRS) with data obtained by conventional X-ray mammography, tissue proteomics, and histopathology in women with breast cancer | At time of breast surgery
  Imaging and spectroscopic studies are performed before surgery. After surgery, this data will be compared and contrast with data obtained from conventional mammograms and the patient's tissue.

SECONDARY OUTCOMES:
Evaluation of the impact of MRS data on treatment planning for radiotherapy and/or surgery in women with breast cancer | After the last scan
  Investigators will evaluate the effectiveness of spectroscopic data used to plan for the patient's post-imaging surgery and/or post-surgical radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Study Chair — Vanderbilt-Ingram Cancer Center